CLINICAL TRIAL: NCT01743274
Title: Does Optical Coherence Tomography Optimise Results of Stenting: The DOCTORS Study
Brief Title: Does Optical Coherence Tomography Optimise Results of Stenting
Acronym: DOCTORS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P/2012/141
Record Dates: First submitted 2012-11-23; First posted 2012-12-06 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Acute Coronary Syndromes
Keywords: acute coronary syndromes; non-ST elevation myocardial infarction; angioplasty; fractional flow reserve; optical coherence tomography
MeSH Terms: conditions — Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Randomization will be performed after initial coronary angiography, once the operator has identified the lesion responsible for the ACS. Patients will be randomly allocated to one of two groups. In the "Control" Group, the angioplasty procedure will be guided by traditional fluoroscopy alone.
  In both groups, fractional flow reserve (FFR) will be measured at the end of the procedure, once the operator considers the result of the angioplasty to be optimal. The average of three consecutive FFR measures will be recorded.
- Optical Coherence Tomography (Experimental): Randomization will be performed after initial coronary angiography, once the operator has identified the lesion responsible for the ACS. Patients will be randomly allocated to one of two groups.
  In the "OCT" group, OCT will be performed to optimise the results of angioplasty. The procedure will be performed according to usual practice, with or without pre-dilation before implantation of one or more stents (drug-eluting or bare metal). In the OCT group, OCT will be performed after initial coronary angiography and at the end of the procedure and the operator will have the possibility to change procedural strategy according to the data immediately available on the OCT images, with the possibility of additional interventions (additional balloon inflations, addition stent implantation, use of GPIIb/IIIa inhibitors and/or thromboaspiration and/or rotational atherectomy).
  Interventions: Procedure: OCT

INTERVENTIONS:
Procedure: OCT — Optical Coherence Tomography (OCT) is a recent imaging modality that yields cross-sectional images with a resolution 10 times greater than that of intravascular ultrasound (IVUS). OCT uses a near-infra-red light source to obtain images of the interior walls of the coronary arteries and is increasingly used to evaluate vulnerable atherosclerotic plaques and assess placement and response to stenting.
  OCT images are acquired by automated pullback over 2 to 3 seconds of the light source that yields a helicoidal image of a longitudinal segment of 50 mm. Intravascular imaging is obtained by injecting contrast medium or saline solution.
  Other Names: Optical coherence tomography
  Arms: Optical Coherence Tomography

SUMMARY:
Optical Coherence Tomography (OCT) is a recent imaging modality that yields cross-sectional images with a resolution 10 times greater than that of intravascular ultrasound (IVUS). OCT uses a near-infra-red light source to obtain images of the interior walls of the coronary arteries and is increasingly used to evaluate vulnerable atherosclerotic plaques and assess placement and response to stenting. - To date, no study has evaluated whether optical coherence tomography (OCT) contributes to optimizing percutaneous coronary intervention (PCI) and stenting.

The DOCTORS study is a randomized, open label study to evaluate whether OCT-guided angioplasty would provide useful clinical information beyond that obtained by angiography, and whether this information would subsequently modify physician behavior and treatment choices. In particular, we will evaluate the impact of changes in procedural strategy resulting from the use of OCT on the value of fractional flow reserve (FFR) obtained after angioplasty and stent implantation of a lesion responsible for non-ST segment elevation acute coronary syndromes.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 to 80 years inclusive, admitted for acute coronary syndrome (ACS) with the following symptoms :

* Clinical signs of ischemia (chest pain) at rest lasting for at least 10 minutes in the previous 72 hours;
* AND at least one of the following two criteria :

  * New ST segment depression ≥1 mm or transitory ST segment elevation (<30 minutes) (≥1 mm) on at least 2 contiguous leads of the ECG; OR
  * Elevation (>upper limit of normal, ULN) of cardiac enzymes (CK-MB, Troponin I or T).

AND Presenting an indication for coronary angioplasty with stent implantation of the target lesion considered to be responsible for the ACS.

AND Written informed consent.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from the study:

* Left main stem disease
* Presence of coronary artery bypass grafts
* Cardiogenic shock or severe hemodynamic instability
* Severely calcified or tortuous arteries
* Persistent ST segment elevation
* One or more other lesions considered angiographically significant and located on the target vessel
* Severe renal insufficiency (creatinine clearance ≤30 mL/min)
* Bacteraemia or septicaemia
* Severe coagulation disorders
* Patients who refuse to sign the informed consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Functional result of the angioplasty procedure as assessed by fractional flow reserve (FFR) | Measured at the end of the angioplasty procedure
  Evaluation of the functional result of the angioplasty procedure as assessed by fractional flow reserve (FFR) at the end of the procedure.
  The average of three consecutive FFR measures will be recorded.

SECONDARY OUTCOMES:
Percentage of patients in whom OCT revealed a sub-optimal result of angioplasty | Assessed during the initial angioplasty procedure (Day 0)
  Assessed by the presence of any one or more of the following criteria:
  Incomplete coverage of the lesion by the stent, Residual stenosis upstream or downstream from the stent, Edge dissection, Presence of thrombus, Tissue protrusion through the stent struts, Stent Malapposition.
Percentage of patients in whom a change in procedural strategy was decided based on the information obtained from OCT images | During the initial angioplasty procedure, as soon as the operator decides whether or not to proceed with additional interventions based on OCT data (Day 0)
  Any one or more of the following criteria based on the information obtained from OCT images:
  Diameter and length of implanted stents Supplementary balloon inflations Implantation of supplementary stent(s) Use of glycoprotein (GP) IIb/IIIa inhibitors Use of thrombo-aspiration Use of rotational atherectomy
Safety of OCT in the context of angioplasty for ACS | At the end of the angioplasty procedure (Day 0) and up to 24 hours (for peak troponin and creatinine clearance)
  Safety as assessed by the following criteria:
  * Duration of the procedure
  * Fluoroscopy time
  * Quantity of contrast medium used
  * Procedural complications (no reflow, coronary perforation, occlusive dissection, spasm, stent occlusion, troponin peak at 24 hours, creatinine clearance at 24 hours)
Adverse cardiac events at 6 months | Recorded by telephone contact with the patient, the treating physician or general practitioner or cardiologist at 6 months after initial angioplasty
  Any one or more of the following:
  * Death
  * Recurrent MI
  * Stent thrombosis
  * Repeat revascularisation of the target vessel
Determination of a threshold value for quantitative OCT measures (i.e. minimal lumen diameter and minimal lumen area) that best predict a fractional flow reserve value >=0.90. | At the end of the initial angioplasty procedure (Day 0)
  Determination of a threshold value for quantitative OCT measures (i.e. minimal lumen diameter and minimal lumen area) that best predict a fractional flow reserve (FFR) value >=0.90.
Identification of quantitative OCT (i.e. minimum lumen diameter and minimum lumen area) variables that predict FFR as measured at the end of the initial angioplasty procedure. | At the end of the initial angioplasty procedure (Day 0)
  Identification of quantitative OCT (i.e. minimum lumen diameter and minimum lumen area) variables that predict the value of fractional flow reserve as measured at the end of the initial angioplasty procedure on day 0.
Comparison between online and offline analyses of OCT data | Analysis of offline data is performed centrally, and comparison will be performed once both online and offline analysis data are performed (Day 90)
  Comparison between results of online and offline analyses of OCT data.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas F. Meneveau, MD, Principal Investigator — University Hospital Besancon, France
Locations (8):
- France (8):
  - Annecy Hospital, Annecy, Metz-Tessy
  - Centre Hospitalier, Belfort
  - University Hospital Jean Minjoz, Besançon
  - Centre Hospitalier de Chambery, Chambéry
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier Universitaire Régional, Lille
  - Institut Mutualiste Montsouris, Paris
  - Nouvel Hôpital Civil, Strasbourg

REFERENCES:
- [Background] Meneveau N, Ecarnot F, Souteyrand G, Motreff P, Caussin C, Van Belle E, Ohlmann P, Morel O, Grentzinger A, Angioi M, Chopard R, Schiele F. Does optical coherence tomography optimize results of stenting? Rationale and study design. Am Heart J. 2014 Aug;168(2):175-81.e1-2. doi: 10.1016/j.ahj.2014.05.007. Epub 2014 May 24. PMID 25066556
- [Result] Meneveau N, Souteyrand G, Motreff P, Caussin C, Amabile N, Ohlmann P, Morel O, Lefrancois Y, Descotes-Genon V, Silvain J, Braik N, Chopard R, Chatot M, Ecarnot F, Tauzin H, Van Belle E, Belle L, Schiele F. Optical Coherence Tomography to Optimize Results of Percutaneous Coronary Intervention in Patients with Non-ST-Elevation Acute Coronary Syndrome: Results of the Multicenter, Randomized DOCTORS Study (Does Optical Coherence Tomography Optimize Results of Stenting). Circulation. 2016 Sep 27;134(13):906-17. doi: 10.1161/CIRCULATIONAHA.116.024393. Epub 2016 Aug 29. PMID 27573032
- [Result] Meneveau N, Ecarnot F. Response by Meneveau and Ecarnot to Letter Regarding Article, "Optical Coherence Tomography to Optimize Results of Percutaneous Coronary Intervention in Patients With Non-ST-Elevation Acute Coronary Syndrome: Results of the Multicenter, Randomized DOCTORS Study (Does Optical Coherence Tomography Optimize Results of Stenting)". Circulation. 2017 Feb 28;135(9):e142-e143. doi: 10.1161/CIRCULATIONAHA.116.026277. No abstract available. PMID 28242645